CLINICAL TRIAL: NCT00244946
Title: Immune Consolidation With Activated T Cells Armed With OKT3 x Rituxan (Anti-CD3 x Anti-CD20) Bispecific Antibody (CD20Bi) After Peripheral Blood Stem Cell Transplant for High Risk CD20+ Non-Hodgkin's Lymphomas
Brief Title: Combination Chemotherapy Followed By Autologous Stem Cell Transplant, and White Blood Cell Infusions in Treating Patients With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lawrence Lum, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000446079; P30CA022453 (NIH); WSU-2007-023; RWMC-0639446
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Lymphoma
Keywords: nodal marginal zone B-cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; splenic marginal zone lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Carmustine; Cytarabine; Etoposide; Melphalan; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous lymphocytes,carmustine,etoposide, melphalan, PBSCT (Experimental): * minus Day 8 ADMIT for Hydration
  * minus Day 7 Carmustine 300 mg/m2 x 1 dose
  * minus Day 6 Etoposide 100 mg/m2 q 12 hr; Cytarabine 100 mg/m2 q 12 hr
  * minus Day 5 Etoposide 100 mg/m2 q 12 hr; Cytarabine 100 mg/m2 q 12 hr
  * minus Day 4 Etoposide 100 mg/m2 q 12 hr; Cytarabine 100 mg/m2 q 12 hr
  * minus Day 3 Etoposide 100 mg/m2 q 12 hr; Cytarabine 100 mg/m2 q 12 hr
  * minus Day 2 Melphalan 140 mg/m2 x 1 dose
  * minus Day 1 Day of Rest
  * Day 0 Transplant
  Interventions: Biological: therapeutic autologous lymphocytes; Drug: carmustine; Drug: cytarabine; Drug: etoposide; Drug: melphalan; Procedure: peripheral blood stem cell transplantation (PBSCT)

INTERVENTIONS:
Biological: therapeutic autologous lymphocytes — Lymphocytes collected by standard apheresis technique either prior to or post stem cell mobilization and collection
Drug: carmustine
Drug: cytarabine
Drug: etoposide
Drug: melphalan
Procedure: peripheral blood stem cell transplantation (PBSCT)

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carmustine, etoposide, cytarabine, and melphalan work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. A peripheral stem cell transplant may be able to replace blood-forming cells that were destroyed by chemotherapy. Giving white blood cells, that have been treated in the laboratory with antibodies, may make the transplant work better. Giving combination chemotherapy followed by an autologous stem cell transplant, and white blood cell infusions may be an effective treatment for non-Hodgkin's lymphoma.

PURPOSE: This phase I trial is studying the side effects and best dose of white blood cell infusions when given together with combination chemotherapy, and autologous stem cell transplant in treating patients with non-Hodgkin's lymphoma that has relapsed, is refractory, or is in remission.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of high-dose combination chemotherapy comprising cyclophosphamide, thiotepa, and carboplatin followed by autologous peripheral blood stem cell transplantation and immunotherapy consolidation therapy comprising anti-CD3 x anti-CD20 bispecific antibody (CD20Bi)-activated T cells (ATC) in patients with non-Hodgkin's lymphoma.
* Determine the maximum tolerated dose of CD20Bi-ATC in patients treated with this regimen.
* Determine whether ATC traffic to tumor sites in select patients treated with this regimen.
* Assess the immune reconstitution of B cells and incidence of infection in patients treated with this regimen.
* Compare relapse rates and overall survival of patients treated with this regimen with historical controls.

OUTLINE: This is a dose-escalation study of activated T cells.

* Peripheral blood stem cell (PBSC) mobilization and collection: Patients receive filgrastim (G-CSF) subcutaneously (SC) once daily for 5 days. They then undergo leukaphereses to collect peripheral blood stem cells (PBSC). Some of the lymphocytes are treated in the laboratory to produce anti-CD3 x anti-CD20 bispecific antibody (CD20Bi)-activated T cells (ATC).
* High-dose chemotherapy and PBSC transplantation: Patients receive carmustine IV on day -7, etoposide IV twice daily and cytarabine IV twice daily on days -6, -5, -4, and -3, and melphalan IV on day -2. Autologous PBSC are reinfused on day 0.
* Immunotherapy consolidation: Patients receive immunotherapy consolidation comprising CD20Bi-ATC IV over 15-30 minutes starting on day 4, once a week for 4 weeks for a total of four infusions.

Cohorts of 3-6 patients receive escalating doses of CD20Bi-ATC until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

After completion of study treatment, patients are followed periodically for survival.

PROJECTED ACCRUAL: A total of 12-24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed CD20+ non-Hodgkin's lymphoma

  * Disease is refractory, relapsed, or in remission
* Measurable or evaluable disease

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Hemoglobin > 8 g/dL
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 50,000/mm^3

Hepatic

* Bilirubin ≤ 2.0 mg/dL
* SGOT or SGPT ≤ 2.5 times normal
* No history of severe hepatic dysfunction

Renal

* Creatinine ≤ 2.0 mg/dL OR
* Creatinine clearance ≥ 60 mL/min
* No uncompensated major adrenal dysfunction
* BUN < 1.5 times normal

Cardiovascular

* No severe cardiac dysfunction
* No major heart disease
* LVEF ≥ 50% by MUGA
* No uncontrolled hypertension
* No congenital or acquired heart disease or cardiac arrhythmias unless cardiac consult and evaluation are done

Pulmonary

* DLCO ≥ 50% of normal
* No symptomatic obstructive or restrictive disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infections
* HIV negative
* No significant skin breakdown from tumor or other diseases
* Dental evaluation and teeth cleaning with no potential sources of infection required
* No uncompensated major thyroid dysfunction

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior stem cell transplantation

Chemotherapy

* No prior total doxorubicin or daunorubicin dose ≥ 450 mg/m^2 unless endomyocardial biopsy shows < grade 2 drug effect AND ejection fraction ≥ 50% by gated blood pool scan

Endocrine therapy

* No concurrent hormonal therapy except steroids for adrenal failure, septic shock, or pulmonary toxicity or hormones for non-disease-related conditions (e.g., insulin for diabetes)

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-03; Primary Completion 2010-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To perform a dose escalation trial of ATC armed with CD20Bi immunotherapy after PBSCT to determine the maximum tolerated dose (MTD) of ATC armed with CD20BI. | When two patienst at any dose levet have their infusion stopped due to side effects.
  This will be the called the maximum tolerated dose. The maximum tolerated dose (MTD) is defined as the dose level below the one at which the side effects are serious enough to prevent an increase in the dose or level of the treatment.

SECONDARY OUTCOMES:
Evaluate the toxicities of ATC infusions armed with CD20Bi | 2 weeks (+/- 7 days), 1, 2, 3, 6 months (+/- 7 days) and 12, and 24 months (+/- one month) after Peripheral Blood Stem Cell Transplants (PBSCT)
Evaluate immune B-cell recovery after ATC infusion | 2 weeks (+/- 7 days), 1, 2, 3, 6 months (+/- 7 days) and 12, and 24 months (+/- one month) after Peripheral Blood Stem Cell Transplants (PBSCT)
Evaluate response rates of infusions and compare relapse rates and overall survival to historical controls | 1, 2, 4, 8, 16 and/or 24, 48 and 72 hours post infusion
  Survival follow-up: 1 year, 3 years, 5 years and 10 years after transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence G. Lum, MD, DSc, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States